CLINICAL TRIAL: NCT07051720
Title: Visual Performance, Patient Satisfaction, and Quality of Vision Outcomes in Presbyopia-Correcting IOLs: A Prospective Clinical Study
Brief Title: Head-to-Head Comparison of Five Enhanced Depth of Focus IOLs and One Monofocal IOL
Acronym: AKA-Reports
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Augenklinik Ahaus G + H GmbH & Co. KG (Other)
Responsible Party: Principal Investigator, Matthias Gerl, CEO, Augenklinik Ahaus G + H GmbH & Co. KG
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-819-f-S
Record Dates: First submitted 2025-06-16; First posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Cataract and IOL Surgery; IOL Implantation; Presbyopia Correction; Extended Depth of Focus
Keywords: Cataract surgery; Extended depth-of-focus; EDOF; Intraocular lens; Presbyopia correction; Spectacle independence; Visual outcomes; Patient satisfaction; TECNIS Eyhance; AcrySof IQ Vivity; LuxSmart; CT Asphina; RayOne EMV; Eyecryl SERT
MeSH Terms: conditions — Cataract; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: This was a prospective, single-center, patient-preference, comparative clinical trial. The participants were provided with comprehensive information regarding each IOL option, including optical principles, expected visual outcomes, potential advantages, and associated limitations. Following detailed counseling and informed consent, patients selected their preferred IOL based on their individual needs, lifestyle requirements, and risk tolerance. The patient-preference design was selected over randomized controlled trial methodology for several considerations: first, to respect patient decision in IOL selection, which is standard practice in premium IOL surgery; second, to minimize ethical concerns associated with randomizing patients to potentially suboptimal treatments based on their individual needs; and third, to provide a real-world evidence regarding patient-chosen outcomes and satisfaction levels.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (6):
- CT ASPHINA 409M IOL group (Experimental): The monofocal intraocular lens CT ASPHINA 409M (Carl Zeiss Meditec AG, Germany) will be implanted during catarct surgery
  Interventions: Device: Bilateral implantation of CT ASPHINA 409M
- TECNIS Eyhance ICB00 IOL group (Experimental): The intraocular lens TECNIS Eyhance ICB00 (Johnson & Johnson Surgical Vision, Irvine, CA, USA) will be implanted during catarct surgery
  Interventions: Device: Bilateral implantation of TECNIS Eyhance ICB00
- AcrySof® IQ Vivity® IOL group (Experimental): The intraocular lens AcrySof® IQ Vivity® (Alcon Laboratories, Fort Worth, TX, USA) will be implanted during catarct surgery
  Interventions: Device: Bilateral implantation of AcrySof® IQ Vivity®
- LuxSmart™ IOL group (Experimental): The intraocular lens LuxSmart™ (Bausch+Lomb, Rochester, NY, USA) will be implanted during catarct surgery
  Interventions: Device: Bilateral implantation of LuxSmart™
- Eyecryl SERT IOL group (Experimental): The intraocular lens Eyecryl SERT (Biotech Healthcare Group, Luzern, Switzerland) will be implanted during catarct surgery
  Interventions: Device: Bilateral implantation of Eyecryl SERT
- RayOne EMV IOL group (Experimental): The intraocular lens RayOne EMV (Rayner Intraocular Lenses Ltd.) will be implanted during catarct surgery
  Interventions: Device: Bilateral implantation of RayOne EMV

INTERVENTIONS:
Device: Bilateral implantation of CT ASPHINA 409M — Patients will be implanted with CT ASPHINA 409M during catarct surgery. The CT Asphina 409M has been commercially available for several years and is widely used in clinical practice. Designed with aberration-neutral optical properties, it could improve contrast sensitivity and visual quality. This monofocal aspheric IOL features four-point plate haptics and a one-piece design made from hydrophilic acrylic material with hydrophobic surface properties. It also has an overall diameter of 11 mm and a 6 mm optical diameter. The lens has a sharp posterior optic edge to minimize posterior capsule opacification. It is ideally suited as a comparative referent lens to new EDOF IOLs.
  Arms: CT ASPHINA 409M IOL group
Device: Bilateral implantation of TECNIS Eyhance ICB00 — Patients will be implanted with TECNIS Eyhance ICB00 during catarct surgery. TECNIS Eyhance ICB00 is a one-piece, posterior chamber lens with an overall diameter of 13.0 mm and an optic diameter of 6.0 mm. The lens has a spherical posterior surface and a modified aspheric anterior surface that offers a smooth and continuous change in power from the periphery to the center of the lens, without a demarcation zone.
  Arms: TECNIS Eyhance ICB00 IOL group
Device: Bilateral implantation of AcrySof® IQ Vivity® — Patients will be implanted with AcrySof® IQ Vivity® during catarct surgery. The AcrySof® IQ Vivity® is a single-piece, hydrophobic acrylic IOL that utilizes non-diffractive wavefront-shaping technology (X-wave™) on its anterior surface to achieve an extended range of vision. Its aspheric anterior surface features a 2.2 mm central zone composed of two smooth transition elements: the first forms a slightly elevated plateau (~1 µm) that stretches the wavefront, while the second shifts the wavefront to create a negative extended focal range. Together, these elements could create advanced and delayed wavefronts resulting in a continuous extended focal range instead of multiple focal points, while optimizing light transmission. This UV-absorbing and blue light filtering foldable IOL has a refractive index of 1.55 at 35 °C, an optic diameter of 6 mm and an overall length of 13 mm. The lens is available in spherical powers ranging from +10.0 to +30.0 diopters.
  Arms: AcrySof® IQ Vivity® IOL group
Device: Bilateral implantation of LuxSmart™ — Patients will be implanted with LuxSmart™ during catarct surgery. The LuxSmart™ intraocular lens is a single-piece, acrylic hydrophobic and aspheric IOL with an overall diameter of 11 mm, an optical diameter of 6 mm, and a 4-point fixation haptic design. This non-diffractive IOL utilizes a technology known as Pure Refractive Optics (PRO), incorporating a 2.0 mm central EDOF zone that combines fourth- and sixth-order spherical aberrations of opposite signs designed to improve perceived depth of focus. The paracentral region, on the other hand, is a transition zone meant to gradually decrease the optic vergence from the center to the monofocal periphery. It has also a 360° continuous square edge on the posterior surface to prevent epithelial lens cells migration and posterior capsule opacification.
  Arms: LuxSmart™ IOL group
Device: Bilateral implantation of Eyecryl SERT — Patients will be implanted with Eyecryl SERT during catarct surgery. EyeCryl-SERT (Biotech) is a new advanced monofocal, single-piece hydrophobic IOL with an aspheric surface, continuous vision from distance to intermediate, spectacle independence for intermediate vision, an extended range of vision: >1.75 D at spectacle plane with visual acuity 0.2 LogMAR or better, an intermediate vision up to 57 cm and a design for fast neural adaptation.
  Arms: Eyecryl SERT IOL group
Device: Bilateral implantation of RayOne EMV — Patients will be implanted with RayOne EMV during catarct surgery. RayOne EMV (Rayner) is a new EDOF lens that has recently emerged in the market. It is a truly non-diffractive, single-piece hydrophilic IOL which does not use light splitting technology like many IOLs which increase depth of focus, resulting in low levels of dysphotopsia, similar to standard monofocal lenses. RayOne EMV is the only patented aspheric IOL that induces controlled positive spherical aberration. Compared to a lens with zero spherical aberration, the carefully controlled positive spherical aberration induced by RayOne EMV spreads light along the visual axis, elongating the focal range from far into intermediate with up to 1.5 D of depth of focus (per lens on the spectacle plane).
  Arms: RayOne EMV IOL group

SUMMARY:
Study Goal

The goal of this clinical trial is to compare how well four different types of artificial lenses (called intraocular lenses or IOLs) help people see after cataract surgery. The main questions it aims to answer are:

Which lens gives the best vision at different distances (far, middle, and close)? How satisfied are patients with their vision after surgery? How often do patients still need glasses after surgery?

Who Can Participate Adults aged 22 to 85 years who need cataract surgery in both eyes and meet specific health requirements.

Study Design

Researchers compared six different lens types:

TECNIS Eyhance - designed to improve middle-distance vision AcrySof IQ Vivity - extends the range of clear vision LuxSmart - uses special optics for better depth of focus Rayner EMV - uses gradual light-bending technology for smooth vision transition Eycryl SERT - modifies light focus to extend clear vision range CT ASPHINA 409M - standard single-focus lens (comparison group)

Participants chose their preferred lens type after learning about each option's benefits and limitations.

What Participants Do? Participants will:

Have cataract surgery on both eyes (1-2 weeks apart) Complete vision tests at multiple distances Take contrast sensitivity tests under different lighting conditions Fill out questionnaires about vision quality and daily activities Attend follow-up visits at 1 day, 1 week, 1 month, and 3 months

This study helps patients and doctors make informed decisions about which type of artificial lens might work best for individual needs and lifestyle.

DETAILED DESCRIPTION:
Study Rationale and Clinical Significance The increasing demand for spectacle independence following cataract surgery has driven the development of advanced intraocular lens (IOL) technologies that extend beyond traditional monofocal designs. This prospective comparative study addresses a critical gap in understanding the real-world performance of contemporary extended depth-of-focus (EDOF) IOLs versus premium monofocal lenses.

Intermediate Vision Focus: Modern lifestyle demands have elevated the importance of intermediate visual function, particularly for distances between 60-80 cm, which encompass critical daily activities including computer work, dashboard viewing, kitchen tasks, and tablet reading. Traditional monofocal IOLs inherently limit functional vision to a single focal distance, necessitating spectacle dependence for intermediate and near visual tasks. This study specifically evaluates how different optical approaches address this intermediate vision gap.

EDOF Technology Principles: The study examines five distinct optical strategies for extending depth of focus: wavefront-shaping technology (AcrySof IQ Vivity), progressive power profiles (TECNIS Eyhance), refractive aberration manipulation (LuxSmart), continuous transition diffractive optics (Rayner EMV), and spherical aberration modulation (Eycryl SERT). Each represents a different approach to creating an elongated focal point rather than discrete foci, theoretically providing enhanced intermediate performance while minimizing visual disturbances associated with multifocal designs.

Study Design and Methodology Design Framework: This prospective, single-center, comparative clinical trial employs a patient-preference methodology rather than traditional randomization. This approach reflects real-world clinical practice where IOL selection involves shared decision-making between surgeon and patient based on individual visual needs, lifestyle requirements, and risk tolerance.

Patient-Preference Rationale: The patient-preference design was selected to: (1) respect patient autonomy in premium IOL selection, (2) minimize ethical concerns associated with randomizing patients to potentially suboptimal treatments based on individual needs, and (3) generate clinically relevant real-world evidence regarding patient-chosen outcomes and satisfaction levels.

Surgical Standardization: All procedures are performed by a single experienced surgeon using standardized phacoemulsification technique with identical surgical parameters: 2.5mm superior corneal incision, 5.5mm continuous curvilinear capsulorhexis, horizontal chop phacoemulsification, and bilateral same-model IOL implantation. Target refraction aims for emmetropia with slight myopic bias.

Primary Assessment Domains Intermediate Visual Performance Distance-Specific Testing: The protocol emphasizes comprehensive intermediate visual assessment at two critical distances: 80cm and 60cm. These distances represent distinct functional zones - 80cm corresponds to automobile dashboard and extended arm's length tasks, while 60cm represents standard computer monitor and kitchen counter distances.

Measurement Methodology: Both uncorrected intermediate visual acuity (UIVA) and distance-corrected intermediate visual acuity (DCIVA) are assessed monocularly and binocularly under standardized photopic conditions (85 cd/m²) using high-contrast charts. Multiple chart sets prevent memorization effects across repeated assessments.

Clinical Significance Threshold: The study is powered to detect clinically meaningful differences of 0.1 logMAR in DCIVA, representing approximately one line of visual acuity improvement that translates to functional benefits for intermediate tasks.

Defocus Curve Analysis Defocus curve: Binocular defocus curve testing employs defocus lenses from +1.50D to -2.50D in randomized order, corresponding to simulated viewing distances from infinity to 40cm.

Depth of Focus Quantification: Two threshold levels (0.1 and 0.2 logMAR) define depth of focus as the dioptric range from 0.00D defocus to the largest negative defocus value maintaining threshold visual acuity. This methodology provides standardized assessment of extended focal range capabilities across IOL technologies.

Functional Vision Range: The defocus curve demonstrates each IOL's usable vision range, identifying optimal performance zones and transition points where visual quality degrades.

Contrast Sensitivity Assessment Multi-Condition Testing: Contrast sensitivity evaluation employs the Functional Vision Analyzer across five spatial frequencies (1.5, 3.0, 6.0, 12.0, and 18.0 cycles per degree) under three standardized lighting conditions: photopic (85 cd/m²), mesopic (3.0 cd/m²), and mesopic-with-glare (3.0 cd/m² background with 28 lux glare source).

Real-World Simulation: The three testing conditions simulate actual visual environments: photopic represents daylight conditions, mesopic simulates twilight or indoor lighting, and mesopic-with-glare replicates challenging scenarios such as night driving with oncoming headlights.

Patient-Reported Outcomes

Validated Questionnaires: Two established instruments assess subjective visual experience:

Visual Function Index-14 (VF-14): Evaluates functional visual performance across 14 daily activities including reading, driving, recognizing faces, and performing fine tasks. Each item scores 0-4 with responses weighted by individual importance, generating a 0-100 scale where higher scores indicate better visual function.

McAlinden's Quality of Vision: Assesses patient-reported visual symptoms including glare, halos, starbursts, hazy vision, distortion, and focusing difficulties. Three Rasch-tested scales measure symptom frequency, severity, and bothersome impact on daily activities.

Spectacle Independence Assessment: Comprehensive evaluation of spectacle dependence across distance, intermediate, and near tasks, with particular emphasis on complete spectacle independence rates and task-specific visual function.

Statistical Methodology Sample Size Calculation: Power analysis targets detection of 0.1 logMAR differences in DCIVA with 90% power and α=0.05, accounting for 10% attrition, requiring 200 eyes (25 patients per group).

Analysis Approach: Generalized linear modeling with inverse Gaussian regression and identity link accommodates logMAR data characteristics.

Multiple Comparison Control: Sequential Bonferroni correction controls Type I error while maintaining statistical power, with the monofocal CT ASPHINA 409M serving as the reference comparator for all pairwise analyses.

Clinical Assessment Timeline Preoperative Evaluation: Comprehensive baseline assessment includes biometry, corneal tomography, specular microscopy, optical coherence tomography, and complete ophthalmologic examination to ensure optimal surgical candidacy and establish baseline parameters.

Postoperative Follow-up: Standardized assessments at 1 day, 1 week, 1 month, and 3 months postoperatively. Primary endpoints are assessed at 1 and 3 months to capture visual stabilization and adaptation effects.

Safety Monitoring: Continuous assessment of IOL stability, posterior capsule opacification development, and complication rates throughout the follow-up period.

Innovation and Clinical Impact This protocol represents the first comprehensive head-to-head comparison of four contemporary IOL technologies using standardized methodology and validated outcome measures. The emphasis on intermediate visual performance, quantitative depth of focus analysis, multi-condition contrast sensitivity assessment, and patient-reported outcomes provides clinically relevant data for evidence-based IOL selection and patient counseling in modern cataract surgery practice.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral implantation of the same intraocular lens (IOL) model
* Expected postoperative best-corrected distance visual acuity (BCDVA) of 0.8 (decimal) or better
* Regular corneal astigmatism less than 1 diopter

Exclusion Criteria:

* Endothelial cell density < 2,000 cells/mm²
* Required IOL power for emmetropia falls outside the available range of +10.0 D to +30.0 D
* Pupillary abnormalities
* Intraocular inflammation
* Recent ocular trauma or ocular surgery that is unresolved/unstable, or which may impair visual outcomes or increase patient risk
* History of corneal refractive surgery (e.g., LASIK, LASEK, PRK)
* Irregular astigmatism, as well as corneal abnormalities or opacities
* Conditions associated with an increased risk of zonular rupture, including capsular or zonular anomalies that may lead to IOL decentration or tilt, such as pseudoexfoliation syndrome, trauma, Marfan syndrome, among others
* Systemic or ocular diseases, or medications, that may impair vision, increase surgical risk, or confound study outcomes
* Clinically significant dry eye disease affecting visual function
* Anticipated need for retinal laser treatment or any other ocular surgical intervention during the study period
* Pregnancy, planned pregnancy, breastfeeding, or any condition associated with hormonal fluctuations that may induce refractive changes
* Continuous contact lens wear within the past 4 weeks
* Inability to understand and/or complete study questionnaires
* Advanced glaucoma with visual field defects
* Age-related macular degeneration (exudative or geographic form)

Ages: 22 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-04-12 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Distance-Corrected Intermediate Visual Acuity at 80cm (Unit: LogMAR) | From enrollment to the end of 3-month follow-up
  Monocular and binocular measurements of distance-corrected intermediate visual acuity (DCIVA) at 80cm in LogMAR.
Distance-Corrected Intermediate Visual Acuity at 60cm (Unit: LogMAR) | From enrollment to the end of 3-month follow-up
  Monocular and binocular measurements of distance-corrected intermediate visual acuity (DCIVA) at 60cm in LogMAR.
Binocular Defocus Curve (Unit: LogMAR) | From enrollment to the end of 3-month follow-up
  Following subjective refraction and determination of BCDVA, binocular defocus curve testing will be performed to evaluate the visual performance by adding defocus lenses from + 1.50 D to - 2.50 D in a randomized order.
BInocular depth of Focus at 0.1 LogMAR threshold (Unit: Diopters) | From enrollment to the end of 3-month follow-up
  In order to comply with the recommendations of the American National Standards Institute (ANSI) Z80.35-2018 guideline regarding the definition of the EDOF IOLs, the binocular depth of focus will be calculated from the binocular defocus curve at 0.1 LogMAR threshold.
Binocular Contrast Sensitivity Function (Unit: Log units) | From enrollment to the end of the 3-month follow-up
  Using the Functional Vision Analyzer (Optec 6500, Stereo Optical Co., Chicago, IL, USA) across five spatial frequencies (1.5, 3.0, 6.0, 12.0, and 18.0 cycles per degree) under three standardized lighting conditions (photopic, mesopic, mesopic with glare).
Vision-related quality of life (Unit: Points on 0-100 scale) | From enrollment to the end of 3-month follow-up
  Using the validated Visual Function Index-14 (VF-14) questionnaire.
Visual symptoms and their impact on daily life (Unit: QoV score 0-100) | From enrollment to the end of 3-month follow-up
  Using the validated McAlinden's Quality of Vision questionnaire.

SECONDARY OUTCOMES:
Corrected distance visual acuity in LogMAR | From enrollment to the end of 3-month follow-up
  Corrected distance visual acuity at 4 m under photopic conditions (approximately 85 cd/m²) in LogMAR.
Distance-corrected near visual acuity in LogMAR | From enrollment to the end of 3-month follow-up
  Distance-corrected near visual acuity (DCNVA) at 40 centimeters in LogMAR.
Endothelial cell density, cells/mm² | From enrollment to the end of 3-month follow-up
  Specular microscopy to measure the endothelial cell density before and after the surgery.
Safety outcomes | From enrollment to the end of 3-month follow-up
  The device-related serious adverse events will be reported.
The development of posterior capsule opacification (PCO) on a scale | From enrollment to the end of 3-month follow-up
  The development of posterior capsule opacification (PCO) and the need for Nd:YAG capsulotomy will be reported as follows:
  1. No PCO.
  2. Peripheral PCO - clinically non-significant.
  3. Clinically significant PCO (affect the visual acuity).
  4. Clinically significant PCO that requires ND:YAG laser capsulotomy.

CONTACTS AND LOCATIONS:
Overall Officials: Labib Alshaweesh, MD, MSc, Study Director — Augenklinik Ahaus; Matthias Müller, Dipl.-Ing.FH, Study Director — Augenklinik Ahaus; dr. med. (Univ. Bud.) Matthias Gerl, MD, Principal Investigator — Augenklinik Ahaus
Locations (1):
- Augenklinik Ahaus, Ahaus, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No